CLINICAL TRIAL: NCT00992407
Title: A Randomized, Open-label, Active-controlled Study to Evaluate Social Functioning of Long Acting Injectable Risperidone and Oral Risperidone in the Treatment of Subjects With Schizophrenia or Schizoaffective Disorder
Brief Title: An Efficacy and Safety Study of Long Acting Injectable Risperidone and Oral Risperidone in Participants With Schizophrenia or Schizoaffective Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR015841; RISSCH4178
Record Dates: First submitted 2009-10-08; First posted 2009-10-09 (Estimated); Results first posted 2014-03-11 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Risperidone; Risperdal
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Risperidone long acting injectables (Experimental)
  Interventions: Drug: Risperidone long acting injectables
- Risperidone tablets (Active Comparator)
  Interventions: Drug: Risperidone tablets

INTERVENTIONS:
Drug: Risperidone long acting injectables — Risperidone long acting injectables will be administered intramuscularly (given into the skin) at a flexible dose of 25, 37.5 or 50 milligram (mg) every 2 weeks up to Week 52. A supplementary oral antipsychotic will also be administered for 3-4 weeks after the initial dose of injection.
  Other Names: Risperdal Consta
  Arms: Risperidone long acting injectables
Drug: Risperidone tablets — Risperidone tablets will be administered orally as 0.5-10 mg daily up to Week 52.
  Other Names: Risperdal
  Arms: Risperidone tablets

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of long acting injectable (LAI) risperidone and oral risperidone treatment on participants with schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions and hallucinations, and withdrawal into the self) or schizoaffective disorder (a mixed psychiatric disorder relating to a complex psychotic state that has features of both schizophrenia and a mood disorder such as bipolar disorder).

DETAILED DESCRIPTION:
This is a randomized (treatment group assigned by chance), open-label (all involved people know the identity of the study drug), active-controlled study to evaluate the improvement in social functioning among participants with schizophrenia taking LAI risperidone and oral risperidone tablet. The study drug will be administered for 52 weeks in flexible dose (range as per Investigator's discretion) and a total of 11 assessment visits will be conducted per participant, including Screening. The participant may be withdrawn from the trial for any medical reason at the sole discretion of the investigator. Before starting the study treatment, participants undergo the period of switching from the previous medication to risperidone for 4 weeks, and then they will be evaluated for tolerability for 2 weeks (run-in period for stabilizing to risperidone). In this 2-week period, participants will take oral risperidone. The efficacy will be primarily evaluated through Personal and Social Performance Scale. Safety will be evaluated through Abnormal Involuntary Movement Scale, Barnes Akathisia Rating Scale, and Simpson-Angus Rating Scale. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria: - Participants who will understand the objectives and necessary procedures of the study and have signed the informed consent form which specified that they were willing to participate in the study - Participants with schizophrenia or schizoaffective disorder requiring long-term antipsychotic drug therapy - Participants with pre-morbid global assessment of functioning score of 71 or higher at Screening - Participants who do not present clinically significant abnormality in biochemistry and electrocardiography - Participants who will be compliant with the study requirements (that is, filling in the questionnaire by themselves) and who are capable of actually performing and willing to implementing them

Exclusion Criteria: - Participants who had taken clozapine for the past three months - Participants with mental retardation (Intelligence Quotient less than 70 at the screening) - Participants with history of or currently with a serious disease (cardiovascular, respiratory, neurological [including seizures or significant cerebrovascular], renal, hepatic, hematologic, endocrine, immunologic or other systemic disease) including clinically relevant abnormal level - Participants who have an allergic or hypersensitive reaction to risperidone or who are unresponsive to risperidone - Pregnant or lactating female participants

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2007-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd. Clinical Trial, Study Director — Janssen Korea, Ltd.
Locations (1):
- Ansan, South Korea

RESULTS

PARTICIPANT FLOW:
Groups:
- Risperidone Injection: Risperidone long acting injectable (LAI) were administered intramuscularly (given into the skin) at a flexible dose of 25, 37.5 or 50 milligram (mg) every 2 weeks up to Week 52.
- Risperidone Tablets: Risperidone tablets were administered orally as 0.5-10 mg daily up to Week 52.
Period: Overall Study
Arm/Group | Risperidone Injection | Risperidone Tablets
Started | 37 | 38
Treated | 20 | 25
Completed | 6 | 14
Not Completed | 31 | 24
Not completed — Protocol Violation | 2 | 1
Not completed — Lost to Follow-up | 3 | 3
Not completed — Adverse Event | 3 | 2
Not completed — protocol Violation & Adverse events | 2 | 4
Not completed — Other | 2 | 0
Not completed — Loss of follow-up & Adverse events | 2 | 1
Not completed — Study medication not administered | 17 | 13

BASELINE CHARACTERISTICS:
Population: "N" (number of participants analyzed) signifies the participants evaluable for this measure.
Groups:
- Total: Total of all reporting groups
Arm/Group | Risperidone Injection | Risperidone Tablets | Total
Number analyzed (Participants) | 17 | 24 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.9 (10.5) | 32.8 (9.4) | 34.5 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 9 | 16 | 25

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Personal and Social Performance (PSP) Scale Score at Week 52
Description: The PSP assesses degree of participant's dysfunction within 4 domains of behavior, socially useful activities, personal and social relationships, self-care, and disturbing and aggressive behavior. The score ranges from 1 to 100, divided into 10 equal intervals to rate degree of difficulty (1=absent to 6=very severe) in each of 4 domains. Based on the 4 domains there will be one total score. Participants with a score of 71 to 100 have a mild degree of difficulty; from 31 to 70, varying degrees of disability; less than or equal to 30, functioning so poorly as to require intensive supervision.
Time Frame: Baseline and Week 52
Population: Intent-to-treat (ITT) population included all randomized participants who received at least one dose of study medication and fulfilled all inclusion and exclusion criteria.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Risperidone Long Acting Injectables: Risperidone long acting injectables were administered intramuscularly (given into the skin) at a flexible dose of 25, 37.5 or 50 milligram (mg) every 2 weeks up to Week 52.
Arm/Group | Risperidone Long Acting Injectables | Risperidone Tablets
Number analyzed (Participants) | 17 | 24
units on a scale
  Baseline | 50.65 (14.19) | 58.71 (9.82)
  Change at Week 52 | 5.35 (9.95) | 5.96 (11.22)
Statistical Analysis 1: Comparison: Risperidone Long Acting Injectables vs Risperidone Tablets; Change from Baseline in Personal and Social Performance (PSP) Scale Score at Week 52; Test type: Non-Inferiority or Equivalence — 80% of power and 0.05 of significance level was used; p = 0.8595, t-test, 2 sided; Mean Difference (Final Values) = -0.61, 95% CI 2-sided [-7.5 to 6.3]

2. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Score at Week 52
Description: The PANSS is a 30-item scale designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor attention, and poor impulse control. The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score consists of the sum of all 30 PANSS items and ranges from 30 to 210. Higher scores indicate worsening.
Time Frame: Baseline and Week 52
Population: ITT population included all randomized participants who received at least one dose of study medication and fulfilled all inclusion and exclusion criteria.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Risperidone Long Acting Injectables | Risperidone Tablets
Number analyzed (Participants) | 17 | 24
units on a scale
  Baseline | 78.0 (11.4) | 69.5 (11.9)
  Change at Week 52 | -11.7 (18.8) | -13.0 (15.7)
Statistical Analysis 1: Comparison: Risperidone Long Acting Injectables vs Risperidone Tablets; Change from Baseline in Positive and Negative Syndrome Scale (PANSS) Score at Week 52; Test type: Non-Inferiority or Equivalence — 80% of power and 0.05 of significance level was used; p = 0.8118, t-test, 2 sided; Mean Difference (Final Values) = 1.29, 95% CI 2-sided [-9.6 to 12.2]

3. Secondary Outcome: Change From Baseline in Clinical Global Impression-Severity Scale (CGI-S) Score at Week 52
Description: The CGI rating scale is a 7-point global assessment that measures the clinician's impression of the severity of illness exhibited by a participant. A rating of 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill participants". Higher scores indicate worsening.
Time Frame: Baseline and Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Risperidone Tablet: Risperidone tablet were administered orally as 0.5-10 mg daily up to Week 52.
Arm/Group | Risperidone Long Acting Injectables | Risperidone Tablet
Number analyzed (Participants) | 17 | 24
units on a scale
  Baseline | 3.4 (1.3) | 2.8 (1.1)
  Change at Week 52 | -0.6 (0.9) | -0.7 (1.1)

4. Secondary Outcome: Change From Baseline in Social Functioning Scale (SFS) Score at Week 52
Description: Social Functioning Scale (SFS) scores from 0 to 223 wherein, following categories were involved: Social Engagement (Score Range 0-15); Interpersonal Communication (Score Range 0-9); Recreational Activities (Score Range 0-45); Social Activities (Score Range 0-66; Independence Competence (Score Range 0-39); Independence Performance (Score Range 0-39); Occupational Activity (Score Range 0-10). Total score is sum of all sub scores and higher score indicates better level of social functioning.
Time Frame: Baseline and Week 52
Population: ITT population included all randomized participants who received at least one dose of study medication & fulfilled eligibility criteria. 'N' (number of participants analyzed) signifies participants evaluable for this measure."n" signifies participants who were evaluated for this measure at specified timepoint for each arm group respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Risperidone Long Acting Injectables | Risperidone Tablets
Number analyzed (Participants) | 16 | 23
units on a scale
  Baseline (n=16, 23) | 99.6 (27.0) | 103.5 (33.2)
  Change at Week 52 (n=4,14) | 2.3 (5.9) | 9.6 (30.2)

5. Secondary Outcome: Change From Baseline in Emotional & Social Functioning Scale (SFS) Score at Week 52
Description: For emotional and SFS, mean scores of neuroticism-extroversion-openness (NEO) personality test, relationship style questionnaire (RSQ), state-trait anger expression inventory (STAXI), positive affect and negative affect schedule (PANAS), emotional intelligence (EI), beck depression inventory (BDI), and beck anxiety inventory (BAI) scales were calculated. Score ranges for each category as:60-300 for NEO, 30-150 for RSQ, 20-80 for STAXI, 20-100 for PANAS, 8-172 for EI, 0-63 for BDI and BAI. Higher score indicates improvement.
Time Frame: Baseline and Week 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Risperidone Long Acting Injectables | Risperidone Tablets
Number analyzed (Participants) | 16 | 21
units on a scale
  NEO personality test: Baseline (n=16,21) | 178.7 (21.8) | 173.7 (22.9)
  EI: Baseline (n=16,21) | 151.4 (23.1) | 152.9 (26.4)
  RSQ: Baseline (n=16,21) | 84.1 (18.9) | 87.1 (14.8)
  STAXI: Baseline (n=16,21) | 37.4 (11.7) | 31.7 (10.8)
  PANAS: Baseline (n=16,21) | 55.1 (14.4) | 51.0 (10.6)
  BDI: Baseline (n=16,21) | 14.8 (11.3) | 16.9 (15.0)
  BAI: Baseline (n=16,21) | 17.9 (16.9) | 15.3 (13.9)
  NEO personality test:Change at Week 52 (n=9,17) | -1.1 (23.8) | 2.2 (21.0)
  RSQ: Change at Week 52 (n=9,17) | -4.1 (16.7) | -8.5 (26.3)
  STAXI:Change at Week 52 (n=9,17) | 0.3 (11.6) | -0.2 (15.6)
  PANAS: Change at Week 52 (n=9,17) | -2.8 (14.2) | -2.8 (17.3)
  EI: Change at Week 52 (n=9,17) | 2.2 (25.5) | 2.4 (19.5)
  BDI:Change at Week 52 (n=9,17) | 1.7 (9.6) | -6.3 (11.1)
  BAI: Change at Week 52 (n=9,17) | 0.9 (12.2) | -3.9 (12.1)

6. Secondary Outcome: Change From Baseline in Verbal Working Memory (VWM) Response Based on Neurocognitive Function Test (NCFT) at Week 52
Description: The NCFT is neuropsychological test which measures psychological functions. The VWM was measured by Korean-Wechsler Adults Intelligence Scale (K-WAIS), which consists of two subscales, the Verbal scale (6 subtests) and the Performance scale (5 subtests). The verbal tests were: information, comprehension, arithmetic, digit span, similarities, and vocabulary. Arithmetic and Digit Span test of Verbal WAIS scales was conducted. Arithmetic test (arithmetic questions were asked orally) involved calculations that measured concentration while manipulating mental mathematical problems. Digit span test (children were asked to repeat the orally given sequences of numbers either as heard or in reverse order) measured attention, concentration, and mental control. Here, mean number of correct responses in limited time period are reported for arithmetic (calculation) and Digit span. Increase in number of correct response indicates improvement.
Time Frame: Baseline and Week 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Correct responses
Arm/Group | Risperidone Long Acting Injectables | Risperidone Tablets
Number analyzed (Participants) | 11 | 15
Correct responses
  VWM (Calculation):Baseline (n=11,14) | 7.5 (2.2) | 9.3 (4.1)
  VWM (Numbers):Baseline (n=11,14) | 11.6 (5.1) | 11.8 (4.6)
  VWM (Calculation):Change at Week 52 (n=7,12) | 2.0 (2.8) | 1.0 (4.1)
  VWM (Numbers):Change at Week 52 (n=7,12) | 1.3 (3.6) | 2.3 (3.1)

7. Secondary Outcome: Change From Baseline in Trail Making Test Based on Neurocognitive Function Test (NCFT) at Week 52
Description: The NCFT is neuropsychological test which measures psychological functions. The Trail Making Test is composed of two Parts, A and B. Part A consists of 25 circles printed on a sheet of paper. Each circle contains a number from 1 to 25. The participant's task is to connect the circles with a pencil line as quickly as possible, beginning with the number 1 and proceeding in numerical sequence. Part B consists of 25 circles numbered from 1 to 13 and lettered from A to L. The task in Part B is to connect the circles, in sequence, alternating between numbers and letters. Here, mean number of seconds are represented required to complete each Part.
Time Frame: Baseline and Week 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Risperidone Long Acting Injectables | Risperidone Tablets
Number analyzed (Participants) | 11 | 15
Seconds
  Trail A Making Test:Baseline (n=11,15) | 52.6 (26.6) | 50.7 (28.9)
  Trail B Making Test:Baseline (n=11,15) | 146.0 (74.2) | 147.3 (118.2)
  Trail A Making Test:Change at Week 52 (n=7,12) | 5.9 (14.9) | -7.8 (10.3)
  Trail B Making Test:Change at Week 52 (n=7,12) | -32.3 (59.3) | -19.5 (37.9)

8. Secondary Outcome: Change From Baseline in Working Memory Based on Neurocognitive Function Test (NCFT) at Week 52
Description: The NCFT is neuropsychological test which measures psychological functions. Working memory was assessed using Controlled Oral Word Association Test (COWAT) which measured verbal fluency and is a sub-test of the multilingual aphasia examination. The COWAT uses the three letter set of C, F, and L to assess phonemic fluency. Individuals are given 1 minute to name as many words as possible beginning with one of the letters. The procedure is then repeated for the remaining two letters. More words indicate improvement.
Time Frame: Baseline and Week 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Words
Arm/Group | Risperidone Long Acting Injectables | Risperidone Tablets
Number analyzed (Participants) | 11 | 15
Words
  WM (Digital Span):Baseline (n=10,12) | 11.6 (4.7) | 14.3 (5.1)
  WM (Coris Block): Baseline (n=8,13) | 10.5 (5.3) | 14.9 (5.2)
  WM (Digital Span):Change at Week 52 (n=6,10) | 1.0 (3.4) | 0.5 (3.0)
  WM (Coris Block): Change at Week 52 (n=5,9) | 4.6 (9.6) | -0.7 (4.7)

9. Secondary Outcome: Change From Baseline in Continuous Performance Task (CPT) Based on Neurocognitive Function Test (NCFT) at Week 52
Description: The NCFT is neuropsychological test which measures psychological functions. The CPT assessed CPT (Omissions) and CPT (Commissions). Omission errors indicate the number of times the target was presented, but the participant did not respond/click the mouse. High omission rates indicate that the participant is either not paying attention (distractibility) to stimuli or has a sluggish response. Commission errors indicate the number of times the participant responded but no target was presented. A fast reaction time and high commission error rate points to difficulties with impulsivity. A slow reaction time with high commission and omission errors indicates inattention in general.
Time Frame: Baseline and Week 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Errors
Arm/Group | Risperidone Long Acting Injectables | Risperidone Tablets
Number analyzed (Participants) | 11 | 15
Errors
  CPT (Omissions):Baseline (n=11,15) | 11.0 (13.5) | 14.2 (34.3)
  CPT (Comissions):Baseline (n=11,15) | 17.4 (37.1) | 29.3 (54.5)
  CPT (Omissions):Change at Week 52 (n=7,12) | 1.6 (17.5) | -12.2 (38.4)
  CPT (Comissions):Change at Week 52 (n=7,12) | -3.9 (4.1) | -0.6 (2.3)

10. Secondary Outcome: Change From Baseline in Theory of Mind (TOM) Scale Score at Week 52
Description: The TOM scale is used to assess the ability of participant to infer other's mental states. It includes recognition that other individuals experience thoughts, feelings, intentions, and desires. It is measured by cartoon task, score ranging from 0-30 and stork task which includes stork task set A (false belief), stork task set B (double bluff, white lie, persuasion, misunderstanding), and physical story, score ranging from 0-12, 0-26 and 0-24 respectively. Higher score indicates improvement.
Time Frame: Baseline and Week 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Risperidone Long Acting Injectables | Risperidone Tablets
Number analyzed (Participants) | 11 | 14
units on a scale
  Cartoon task:Baseline (n=11,13) | 13.8 (8.7) | 18.5 (9.3)
  Stork Task Set A: Baseline (n=9,12) | 6.0 (2.0) | 6.6 (2.8)
  Stork Task Set B: Baseline (n=11,14) | 14.2 (6.2) | 15.5 (6.8)
  Cartoon task:Change at Week 52(n=7,11) | 5.0 (7.9) | 2.7 (3.9)
  Stork Task Set A:Change at Week 52(n=7,11) | 1.0 (3.6) | 0.8 (4.8)
  Stork Task Set B:Change at Week 52(n=4,8) | 1.0 (8.3) | 1.5 (3.6)
  Physical story: Baseline (n=11,14) | 12.0 (5.0) | 13.6 (4.4)
  Physical story:Change at Week 52(n=7,11) | 1.4 (5.2) | 2.1 (3.9)

11. Secondary Outcome: Change From Baseline in Psychosocial Well-being Index (PWI) Score at Week 52
Description: Psychosocial Well-being Index (PWI) is a questionnaire about how the participant feels and how the things had been going with them. Total score ranges from 0 to 135, where lower score indicates worsening.
Time Frame: Baseline and Week 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Risperidone Long Acting Injectables | Risperidone Tablets
Number analyzed (Participants) | 16 | 22
units on a scale
  Baseline (n=16,22) | 93.8 (21.9) | 96.0 (14.2)
  Change at Week 52 (n=9,18) | 10.7 (22.1) | 0.7 (15.1)
Statistical Analysis 1: Comparison: Risperidone Long Acting Injectables vs Risperidone Tablets; Change from Baseline in Psychosocial Well-being Index (PWI) Score at Week 52; Test type: Non-Inferiority or Equivalence — 80% of power and 0.05 of significance level was used; p = 0.1768, Student's t-test; Mean Difference (Final Values) = 10.00, 95% CI 2-sided [-4.8 to 24.8]

12. Secondary Outcome: Change From Baseline in Global Assessment of Functioning (GAF) Test Score at Week 52
Description: The GAF is a 100-point tool rating overall psychological, social and occupational functioning of adults. The higher score range (91 to 100) refers to a superior functioning in a wide range of activities, and absence of symptoms. The lower score range (1 to 10) refers to persistent danger of severely hurting self or others; or persistent inability to maintain minimum personal hygiene; or serious suicidal act with clear expectation of death.
Time Frame: Baseline and Week 52
Population: ITT population included all randomized participants who received at least one dose of study medication and fulfilled all inclusion and exclusion criteria. "n" signifies those participants who were evaluated for this measure at the specified time point for each arm group respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Risperidone Long Acting Injectables | Risperidone Tablets
Number analyzed (Participants) | 17 | 24
units on a scale
  Baseline (n=17,24) | 58.3 (16.7) | 63.4 (10.5)
  Change at Week 52 (n=8,17) | 5.4 (11.2) | 5.7 (15.2)
Statistical Analysis 1: Comparison: Risperidone Long Acting Injectables vs Risperidone Tablets; Test type: Non-Inferiority or Equivalence — 80% of power and 0.05 of significance level was used; p = 0.9569, Student's t-test; Mean Difference (Final Values) = -0.33, 95% CI 2-sided [-12.8 to 12.2]

13. Secondary Outcome: Change From Baseline in Scale to Assess Unawareness of Mental Disorder (SUMD) Score at Week 52
Description: The SUMD scale is a semi-structured scale that assesses participant's awareness of and insight into their illness, that is, the present level of insight. SUMD total score ranges from 0-27, with higher scores indicating poorer insight. The scale consists of nine items score ranging from 1 to 3, with higher scores indicating poorer insight. Score for each item is summed to produce the total score.
Time Frame: Baseline and Week 52
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Risperidone Long Acting Injectables | Risperidone Tablets
Number analyzed (Participants) | 17 | 24
units on a scale
  Baseline (n=17,24) | 12.1 (5.1) | 10.6 (5.0)
  Change at Week 52 (n=6,17) | -4.8 (6.2) | -3.5 (3.5)
Statistical Analysis 1: Comparison: Risperidone Long Acting Injectables vs Risperidone Tablets; Test type: Non-Inferiority or Equivalence — 80% of power and 0.05 of significance level was used; p = 0.5294, t-test, 2 sided; Mean Difference (Final Values) = 0.58, 95% CI 2-sided [-5.5 to 2.9]

14. Secondary Outcome: Change From Baseline in Drug Attitude Inventory-10 (DAI-10) Score at Week 52
Description: The DAI-10 is a 10-item questionnaire to assess 1) subjective experience of drug and 2) attitudes and beliefs toward neuroleptics which may influence compliance in schizophrenia participants. Score ranges from (-) 10 to 10. It is the binary scale assessing the participant's subjective response. A 'compliant' response is scored as +1; a dysphoric response is scored as -1. A positive sum of items indicates a positive subjective response (SR); a negative sum of scores indicates a negative SR (non-compliant).
Time Frame: Baseline and Week 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Risperidone Tablet: Risperidone tablets were administered orally as 0.5-10 mg daily up to Week 52.
Arm/Group | Risperidone Injection | Risperidone Tablet
Number analyzed (Participants) | 15 | 18
units on a scale
  Baseline (n=15,18) | 4.1 (4.6) | 5.0 (4.1)
  Change at Week 52 (n=7,15) | -4.7 (7.8) | -1.1 (5.9)

15. Secondary Outcome: Change From Baseline in Members for Outpatients, Members Visiting Inpatients, Affected Members and Visiting Inpatients at Week 52
Description: Healthcare economics questionnaire consists of 13-Questions, which measured disease burden on participant; out of which 4 questions are related to number of members for outpatients, number of members visiting inpatients, number of affected members and number of visiting inpatients. Mean-calculations were done for all questions. Higher value indicates more disease burden. Change from Baseline is the value at Week 52 minus value at Baseline.
Time Frame: Baseline and Week 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: participants
Arm/Group | Risperidone Long Acting Injectables | Risperidone Tablets
Number analyzed (Participants) | 13 | 16
participants
  Members for outpatients:Baseline(n=13,16) | 0.8 (0.4) | 0.7 (0.7)
  Members visiting inpatients (MVI):Baseline(n=6,9) | 2.2 (2.1) | 2.9 (2.6)
  Affected members:Baseline(n=11,14) | 0.6 (0.7) | 0.7 (1.0)
  Visiting inpatients:Baseline(n=7,8) | 6.0 (6.6) | 6.1 (4.6)
  Members for outpatients:Change at Week 52(n=8,13) | -0.3 (0.5) | -0.3 (0.6)
  MVI:Change at Week52(n=0,3) | 0 (0) | -2.7 (3.1)
  Affected members:Change at Week52(n=4,10) | -0.3 (0.5) | -0.4 (0.7)
  Visiting inpatients:Change at Week52(n=0,3) | 0 (0) | -5.0 (5.0)

16. Secondary Outcome: Change From Baseline in Days of Hospitalization, Number of Days Affected by Participants and Family, at Week 52
Description: Healthcare economics questionnaire consists of 13-Questions, which measured disease burden on participant; out of which 3 questions are related to days of hospitalization, number of days affected by participants and family per participant within reporting interval score. Mean-calculations were done for all questions. Change from Baseline is the value at Week 52 minus value at Baseline.
Time Frame: Baseline and Week 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Risperidone Long Acting Injectables | Risperidone Tablets
Number analyzed (Participants) | 11 | 18
days
  Hospitalization days:Baseline(n=11,18) | 19.4 (21.3) | 9.8 (13.4)
  Days affected:Baseline(n=8,11) | 34.0 (46.4) | 24.3 (34.5)
  Family affected days:Baseline(n=9,12) | 2.9 (4.8) | 2.0 (3.4)
  Hospitalization days:Change at Week 52(n=3,12) | -14.0 (24.2) | -10.0 (15.0)
  Days affected:Change at Week 52(n=3,10) | -30.0 (52.0) | -25.3 (33.1)
  Family affected days:Change at Week 52(n=4,10) | -0.3 (2.1) | -1.5 (3.2)

17. Secondary Outcome: Change From Baseline in Total Outpatients and Inpatients Hours at Week 52
Description: Healthcare economics questionnaire consists of 13-Questions, which measured disease burden on participant; out of which 2 questions are related to total outpatients and inpatients hours. Total outpatients hours and total inpatient hours indicate the total hours spent by outpatients and inpatients respectively at Investigator site.Mean-calculations were done for all questions. Higher value indicates more disease burden. Change from Baseline is the value at Week 52 minus value at Baseline.
Time Frame: Baseline and Week 52
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Risperidone Long Acting Injectables | Risperidone Tablets
Number analyzed (Participants) | 9 | 13
hours
  Total outpatients hours:Baseline(n=9,13) | 1.7 (1.0) | 1.6 (0.7)
  Total inpatient hours:Baseline(n=5,8) | 1.4 (1.5) | 1.4 (0.9)
  Total outpatients hours:Change at Week 52(n=4,9) | 0.1 (1.0) | -0.2 (0.4)
  Total inpatient hours:Change at Week 52(n=0,3) | 0.0 (0.0) | -1.0 (1.0)

18. Secondary Outcome: Change From Baseline in Travelling Fee for Outpatients, Hospitalization Travelling Fee and Salary Paid a Participant Before Being Ill at Week 52
Description: Healthcare economics questionnaire consists of 13-Questions, which measured disease burden on participant; out of which 3 questions are related to travelling fee for outpatients, hospitalization travelling fee and salary paid a participant before being ill. Mean-calculations were done for all questions. Travelling fee, hospitalization travelling fee and salary paid were assessed for every past three months. Higher value indicates more disease burden. Change from Baseline is the value at Week 52 minus value at Baseline.
Time Frame: Baseline and Week 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Won
Arm/Group | Risperidone Long Acting Injectables | Risperidone Tablets
Number analyzed (Participants) | 12 | 14
Won
  Travel fee for outpatient(TFO):Baseline(n=12,14) | 4645.8 (4739.6) | 4850.0 (6401.1)
  Hospitalization fee:Baseline(n=4,6) | 3500.0 (4725.8) | 9500.0 (8043.6)
  Salary paid:Baseline(n=4,6) | 0.0 (0.0) | 3000.0 (7348.5)
  TFO:Change at Week 52(n=12,14) | -658.3 (2168.0) | 183.3 (10837.4)
  Hospitalization fee:Change at Week 52(n=0,3) | 0 (0.0) | -7333.3 (9451.6)
  Salary paid:Change at Week 52(n=3,6) | 0 (0.0) | -3000.0 (7348.5)

19. Secondary Outcome: Change From Baseline in Number of Outpatient Clinic Visits at Week 52
Description: Healthcare economics questionnaire consists of 13-Questions, which measured disease burden on participant; out of which 1 question is related to number of outpatient clinic visits. Mean-calculations were done for all questions. Higher value indicates more disease burden. Change from Baseline is the value at Week 52 minus value at Baseline.
Time Frame: Baseline and Week 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: number of visits
Arm/Group | Risperidone Long Acting Injectables | Risperidone Tablets
Number analyzed (Participants) | 13 | 20
number of visits
  Outpatient clinic visits:Baseline(n=13,20) | 4.7 (4.2) | 4.4 (2.5)
  Outpatient clinic visits:Change at Week 52(n=7,14) | 2.4 (6.3) | 1.1 (3.1)

20. Secondary Outcome: Change From Baseline in Abnormal Involuntary Movement Scale (AIMS) Score at Week 52
Description: The AIMS rates the severity of involuntary movements from 0 (none) to 4 (severe), including facial and oral movements, extremity movements, trunk movements, global and judgments, and 2 additional items concerning dental status (yes/no). A total score (ranging from 0 to 28) will be calculated as the sum of items 1 to 7.
Time Frame: Baseline and Week 52
Population: Safety analysis population included all randomized subjects who received risperidone injection or risperidone tablets at least once. "n" signifies those participants who were evaluated for this measure at the specified time point for each arm group respectively.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Risperidone Long Acting Injectables | Risperidone Tablets
Number analyzed (Participants) | 20 | 25
units on a scale
  Baseline (n=20,25) | 0 (4.6) [0 to 3] | 0 (4.1) [0 to 1]
  Change at Week 52 (n=19,20) | 0 (5.6) [-2 to 1] | 0 (4.8) [-1 to 0]

21. Secondary Outcome: Change From Baseline in Simpson and Angus Rating Scale (SAS) Score at Week 52
Description: The SAS rates 10 items from 0 (normal) to 4 (extreme), including gait, arm dropping, shoulder shaking, elbow rigidity, wrist rigidity, leg pendulousness, head rotation, Glabellar tap, tremor and salivation. The SAS global score is the average score (total sum of items score divided by the number of items) and ranges between 0 and 4, where the higher score denotes more severe condition of extra pyramidal symptoms.
Time Frame: Baseline and Week 52
Population: as for outcome 20
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Risperidone Long Acting Injectables | Risperidone Tablets
Number analyzed (Participants) | 20 | 25
units on a scale
  Baseline (n=20,25) | 0 (4.6) [0 to 1] | 0 (4.1) [0 to 0]
  Change at Week 52 (n=19,22) | 0 (5.6) [0 to 0] | 0 (4.8) [0 to 0]

22. Secondary Outcome: Change From Baseline in Barnes Akathisia Rating Scale (BARS) Score at Week 52
Description: The BARS includes an objective rating, 2 subjective ratings of symptoms of akathisia (awareness of restlessness and reported distress related to restlessness: ranging from 0 to 3), and a global clinical rating of akathisia (GCRA), ranging from 0 (absent) to 5 (severe). The global rating score, that is scored separately, is the most relevant measure of severity of akathisia. Higher scores denote worsening akathisia.
Time Frame: Baseline and Week 52
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Risperidone Long Acting Injectables | Risperidone Tablets
Number analyzed (Participants) | 20 | 25
Units on a scale
  Restlessness total score: Baseline(n=20,25) | 0.80 (1.11) | 0.40 (0.71)
  GCRA: Baseline(n=20,25) | 0.40 (0.60) | 0.32 (0.48)
  Restlessness total score:Change at Week52(n=19,22) | -0.16 (1.12) | 0.00 (0.87)
  GCRA: Change at Week 52(n=19,22) | 0.05 (0.71) | -0.09 (0.68)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 52
Description: An adverse event is any untoward medical occurrence in a clinical study participant administered with study treatment. It can be any unfavorable and unintended sign/abnormal finding, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Arm/Group | Risperidone Injection | Risperidone Tablets
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/25
Other Adverse Events (participants affected / at risk) | 11/20 | 13/25
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Risperidone Injection (N=20) | Risperidone Tablets (N=25)
Akathisisa (Nervous system disorders) | 2 (6) | 4 (20)
dystonia (Nervous system disorders) | 1 (1) | 2 (4)
sedation (Nervous system disorders) | 0 (0) | 1 (1)
dysarthria (Nervous system disorders) | 1 (2) | 1 (6)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
headache (Nervous system disorders) | 0 (0) | 1 (1)
Hypersomnia (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1)
Dysphemia (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Obsessive thoughts (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Weight increased (Investigations) | 2 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Amenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less